CLINICAL TRIAL: NCT04889196
Title: The Efficiency and Gingival Health Status of Hall Versus SDF Techniques in the Management of Carious Primary Molars: Randomized Clinical Trial
Brief Title: The Efficiency and Gingival Health Status of Hall Versus SDF Techniques in the Management of Carious Primary Molars
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarah Abdalla Ibrahim Abdalla (Other)
Responsible Party: Sponsor-Investigator, Sarah Abdalla Ibrahim Abdalla, principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120
Record Dates: First submitted 2021-05-01; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The group that have caries in primary molars and treat them with hall technique
  Interventions: Device: hall technique
- experimental group (Experimental): the group that have caries in primary molars and treat them with silver diamine fluoride (SDF) solution would exert a prevention result in managing early childhood caries ECC
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — Previous studies have recommended that Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. the objective is useful in arresting early childhood caries (ECC)
  Arms: experimental group
Device: hall technique — The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method.
  Arms: control group

SUMMARY:
PICO question:

In Comparison to the hall technique , will silver diamine fluoride have equalvent gingival health status in treatment of carious primary molars?

population: children suffering from caries . intervention : silver diamine fluoride. comparison: hall technique outcome:

Primary outcome:

Gingival health measurement device modified gingival index, measurement unit score(0-1-2)

Secondary outcomes:

1. Oral hygiene measurement device modified plaque index , measurement unit score (0-1-2)
2. Time of Treatment measurement device digital chronometer, measurement unit minutes

DETAILED DESCRIPTION:
Dental caries, also known as tooth decay, it can occur in primary teeth in early childhood, is formed through interaction between acid-producing bacteria and carbohydrate. The caries develops in both the crowns and roots of teeth. Progress of caries depended on the lifestyle of the child (as high numbers of cariogenic bacteria, inadequate salivary flow, insufficient fluoride exposure and poor oral hygiene). To avoid this disease should follow the proper oral hygiene and improve lifestyle . A lot of methods found to treatment the decayed tooth - like; Hall technique and Silver diamine fluoride The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method

Previous studies have recommended that Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. the objective is useful in arresting early childhood caries (ECC)

ELIGIBILITY:
Inclusion Criteria:

* Age: From 4 to 6 years
* Clinical diagnosis of tooth with caries in primary molars within enamel or dentin without pulp disease

Exclusion Criteria:

* Tooth with signs and symptoms of pulp necrosis
* Tooth with Root caries
* Tooth with Spontaneous pain

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Gingival health | up to 1 day
  Modified Gingival index (0 = no swelling
  1. = mild swelling, no bleeding after gentle probing
  2. = moderate to severe gingival swelling, bleeding after air drying
Gingival health | at 3 months
  Modified Gingival index (0 = no swelling
  1. = mild swelling, no bleeding after gentle probing
  2. = moderate to severe gingival swelling, bleeding after air drying
Gingival health | at 6 months
  Modified Gingival index (0 = no swelling
  1. = mild swelling, no bleeding after gentle probing
  2. = moderate to severe gingival swelling, bleeding after air drying

SECONDARY OUTCOMES:
Oral hygiene | up to one day
  Modified Plaque index(0 = no plaque
  1. = thin visible plaque, difficult to identify
  2. = thick visible plaque, easily detected
Oral hygiene | at 3 months
  Modified Plaque index(0 = no plaque
  1. = thin visible plaque, difficult to identify
  2. = thick visible plaque, easily detected
Oral hygiene | at 6 months
  Modified Plaque index (0 = no plaque
  1. = thin visible plaque, difficult to identify
  2. = thick visible plaque, easily detected
Treatment time | during procedure
  Digital chronometer
Treatment time | during procedure in the second application at 6 monthes
  Digital chronometer

CONTACTS AND LOCATIONS:
Overall Officials: sherif B Eltaeil, Prof, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elamin F, Abdelazeem N, Salah I, Mirghani Y, Wong F. A randomized clinical trial comparing Hall vs conventional technique in placing preformed metal crowns from Sudan. PLoS One. 2019 Jun 3;14(6):e0217740. doi: 10.1371/journal.pone.0217740. eCollection 2019. PMID 31158253
- See also: A randomized clinical trial comparing Hall vs conventional technique in placing preformed metal crowns from Sudan. — https://pubmed.ncbi.nlm.nih.gov/31158253/